CLINICAL TRIAL: NCT00330902
Title: Randomized Trial of Sulfadoxine-Pyrimethamine Plus Artesunate (SP+AS) Versus SP+AS Plus Primaquine for Clearance of Low Density P. Falciparum Infection in Eastern Sudan
Brief Title: Randomized Trial of Two Antimalarial Treatments for Clearing Low Density P.Falciparum Parasitaemia in Sudan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Tropical Medicine Research Institute (Other); World Health Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGS64
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Plasmodium Infections
Keywords: malaria; subpatent parasitaemia; dry season; primaquine; Plasmodium falciparum infection detected by PCR
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Sulfadoxine pyrimethamine plus three daily doses of artesunate
  Interventions: Drug: sulfadoxine-pyrimethamine (SP) plus artesunate (AS)
- 2 (Experimental): Sulfadoxine pyrimethamine plus artesunate plus primaquine
  Interventions: Drug: primaquine (PQ) plus SP+AS

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine (SP) plus artesunate (AS) — sulfadoxine-pyrimethamine (SP) plus three daily doses of artesunate (AS)
  Arms: 1
Drug: primaquine (PQ) plus SP+AS — single dose of primaquine on day 4
  Arms: 2

SUMMARY:
In areas of seasonal malaria transmission, treatment of carriers of malaria parasites, whose parasitaemia persists at very low levels throughout the dry season, could be a useful strategy for malaria control in areas with a short transmission season. We did a randomized trial to compare two regimens for clearance of low level parasitaemia in the dry season.

DETAILED DESCRIPTION:
104 individuals with low density Plasmodium falciparum infection detected by polymerase chain reaction (PCR) were randomized to receive sulfadoxine-pyrimethamine and three daily doses of artesunate (SP+AS) or SP+AS and a dose of primaquine (SP+AS+PQ), and were followed up for 14 days during the transmission-free season in Eastern Sudan. Subjects were visited on days 3, 7 and 14 after the start of treatment to record any adverse events and to detect P.falciparum using PCR. PCR positive samples were tested for gametocytes using RT-PCR. Packed cell volume was measured on days 7 and 14.

ELIGIBILITY:
Inclusion Criteria:

* infection with P.falciparum detected by PCR

Exclusion Criteria:

* pregnancy
* severe anaemia
* fever or other signs of illness
* history of allergy to sulfa drugs
* presence of other species of Plasmodium detected by microscopy

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2004-01; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
P.falciparum parasitaemia detected by PCR on days 3,7 and 14. | 14 days from start of treatment

SECONDARY OUTCOMES:
Presence of gametocytes detected by RT-PCR on days 3, 7 and 14. | 14 days from start of treatment
Packed Cell volume on days 7 and 14. | Over 14 days from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Badria B El Sayed, PhD, Principal Investigator — TMRI, Khartoum; Omer Z Baraka, MD, Study Chair — Faculty of Medicine, University of Khartoum
Locations (1):
- Tropical Medicine Research Institute, Khartoum, Sudan

REFERENCES:
- [Derived] El-Sayed B, El-Zaki SE, Babiker H, Gadalla N, Ageep T, Mansour F, Baraka O, Milligan P, Babiker A. A randomized open-label trial of artesunate- sulfadoxine-pyrimethamine with or without primaquine for elimination of sub-microscopic P. falciparum parasitaemia and gametocyte carriage in eastern Sudan. PLoS One. 2007 Dec 12;2(12):e1311. doi: 10.1371/journal.pone.0001311. PMID 18074034